CLINICAL TRIAL: NCT03453736
Title: A Qualitative Study of Staff Experiences and Practices Within the Robotic Theatre Setup
Brief Title: Staff Experiences in Robotic Theatres
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0647; 237227 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2018-02-19; First posted 2018-03-05 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Robotic Staff Experiences
Keywords: Robotic surgery; theatre staff; teamwork; patient safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic procedures: Experiences and practices in Robotic theatres will be studied via semi-structured interviews with staff as well as team observations during real time robotic surgery. As the study is a qualitative one, data collection will continue till we reach saturation of theoretical categories. We expect 20 interviews and 10 observations to suffice.
  Interventions: Other: No intervention
- Non-Robotic procedures: Staff involved in robotic surgery will have almost definitely worked in non-robotic theatres ie major abdominal and laparoscopic. Staff interviews will explore differences in experiences and practices between these different theatre setups.
  In addition, we aim to observe further 5 non-robotic procedures to evaluate staff teamwork and communication within the more regular theatre setup.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a qualitative study involving staff interviews and observations. No intervention is being applied.

SUMMARY:
Studies have shown that team work impacts patients safety. This is particularly the case in surgical theatres where individuals from different backgrounds (surgeon, anaesthetists, nurses, ..etc) work together to achieve a common goal which is looking after the patient. The robotic theatre set up is different due to the physical separation of the surgeon from the patient and the rest of the team. This may represent a communication challenge. The Study investigators aim to study theatre staff experiences and practices of communication and teamwork in this special setup, investigating any challenges participants may be facing and possible ways of adapting to them. Staff opinions and suggestions for improvement will be explored for utmost surgical performance and patient safety.

The study will involve two parts:1) individual staff interviews and 2) teamwork observations during real life surgery. The two parts should complement each other giving an overall picture of the teamwork in the robotic theatre setup.

ELIGIBILITY:
Inclusion Criteria:

1. Robotic theatre staff as above.
2. Willing and able to participate.
3. Good command of the English language.

Exclusion Criteria:

1. Theatre staff not involved in robotic surgery.
2. Participants not willing / unable to participate.
3. Staff that have not worked in a conventional theatre setup before.
4. Inability to read/speak/understand English.
5. Lack of capacity for consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be theatre staff, from any surgical discipline, who are involved in robotic surgery practice at University Hospitals of Leicester and Cambridge University Hospital. This includes, but not limited to surgeons (primary and assistants), nurses (scrub, circulating, or student), anaesthetists (including trainees) and operating department practitioners (ODP).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Robotic staff experiences. | 1 year
  This will be explored using individual interviews and team observations. Textual data of interview transcripts and observation field notes will be analysed using constant comparative method.
Robotic staff practices | 1 year
  This will be explored using individual interviews and team observations. Textual data of interview transcripts and observation field notes will be analysed using constant comparative method.

SECONDARY OUTCOMES:
Staff communication in robotic theatres. | 1 year
  This will be explored using individual interviews and team observations. Textual data of interview transcripts and observation field notes will be analysed using constant comparative method.
Staff teamwork | 1 year
  This will be explored using individual interviews and team observations. Textual data of interview transcripts and observation field notes will be analysed using constant comparative method.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No